CLINICAL TRIAL: NCT05793957
Title: Anxiety in the Context of Chemotherapy Infusion: Is There an Association Between the Use of Virtual Reality Goggles and Changes in Anxiety-Related Symptoms?
Brief Title: Use of Virtual Reality Goggles During Chemotherapy Infusion to Reduce Anxiety-Related Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ryan Li, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00025461; NCI-2023-01954 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00025461 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2023-03-17; First posted 2023-03-31 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Breast Neoplasm; Malignant Head and Neck Neoplasm; Malignant Solid Neoplasm; Malignant Thoracic Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (VR) (Experimental): Patients use VR during chemotherapy infusion on study.
  Interventions: Other: Questionnaire Administration; Other: Virtual Technology Intervention
- Group 2 (Smartphone) (Active Comparator): Patients use smartphone during chemotherapy infusion on study.
  Interventions: Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Use smartphone
  Arms: Group 2 (Smartphone)
Other: Virtual Technology Intervention — Use VR headset
  Other Names: Virtual Reality Intervention; Virtual Technology
  Arms: Group 1 (VR)

SUMMARY:
This clinical trial evaluates the use of virtual reality (VR) goggles during chemotherapy infusion to reduce anxiety-related symptoms in patients with head and neck, thoracic, hematologic, and breast cancers. Virtual reality headsets provide the ability for users to explore a simulated, three-dimensional environment with which users can interact. In virtual reality users can play interactive games, enjoy relaxing experiences, and watch immersive videos. The use of VR goggles may help with anxiety management during chemotherapy infusion.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effectiveness of VR therapy in reducing severity of anxiety symptoms during chemotherapy infusion, compared to participants utilizing a smartphone as a control.

SECONDARY OBJECTIVES:

I. To evaluate whether there is a short-term effect of VR use in anxiety levels.

II. To assess participant satisfaction with their chemotherapy infusion experience in the control and treatment groups.

EXPLORATORY OBJECTIVE:

I. To assess participants' reported adverse effects associated with VR headset use.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP 1: Patients use VR during chemotherapy infusion on study.

GROUP 2: Patients use smartphone during chemotherapy infusion on study.

ELIGIBILITY:
Inclusion Criteria:

* English speaking: Ability to interact with virtual reality content may be impacted by inability to understand English; moreover, paper questionnaires will only be provided in English.
* Older than 18 years of age, and younger than 89 years of age. All sexes/gender identities and members of all races and ethnic groups will be included.
* Planned to receive chemotherapy infusion for head and neck, breast, thoracic, and hematologic cancers at the Oregon Health & Science University (OHSU) South Waterfront Center for Health & Healing building 2 (there are no restrictions related to prior chemotherapy infusions or other cancer treatments).
* Chemotherapy treatment lasting at least 10 minutes.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Social or psychiatric conditions that may interfere with compliance.
* Reconstruction, incisions, wounds, wound care, or injury that impact the ability to place on the VR headset. This would limit the ability to utilize the VR headset.
* History of seizure or epilepsy.
* History of vertigo or persistent dizziness.
* Use of cardiac pacemaker, requirement for hearing aid on at all times, or have defibrillators.
* Children.
* Pregnant women.
* Decisionally impaired adults.
* Prisoners.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Difference in anxiety levels | Before the start of chemotherapy infusion and 30-minutes of virtual reality (VR)/smartphone use is completed
  Will be assessed in the treatment and control groups determined by the difference in the scores provided by the State Anxiety Inventory before and right after VR use. Range of scores is 20-80, the higher score indicating greater anxiety. Will be compared using two-sample t-test to compare the anxiety levels change before and after VR between intervention group and control group (VR vs control). The effect of VR on anxiety levels will be described using a linear regression model addressing the unanticipated imbalance between treatment groups after randomization adjusting for the confounder.

SECONDARY OUTCOMES:
Short-term difference in anxiety levels | Before VR goggle use and immediately after chemotherapy infusion is complete
  Will be assessed by the difference in anxiety levels right before VR use and immediately after chemotherapy infusion is completed as provided by the State Anxiety Inventory using a two sample t-test. Range of scores is 20-80, with a higher score indicating greater anxiety.
Participants' satisfaction with the VR device | Immediately after chemotherapy infusion is complete
  Will be assessed by an investigator-designed satisfaction questionnaire after chemotherapy completion to assess participants' satisfaction with the VR device using descriptive statistics to summarize this data.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Li, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States